CLINICAL TRIAL: NCT00003750
Title: A Phase I/IB Intergroup Trial of the HU14.18-IL2 Fusion Protein in Children With Refractory Neuroblastoma and Other GD2 Positive Tumors
Brief Title: Biological Therapy in Treating Children With Refractory or Recurrent Neuroblastoma or Other Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL0018; COG-ADVL0018 (Other: Children's Oncology Group); CDR0000066870 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Melanoma (Skin); Neuroblastoma; Sarcoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: metastatic osteosarcoma; recurrent neuroblastoma; recurrent osteosarcoma; recurrent melanoma; unspecified childhood solid tumor, protocol specific; metastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma
MeSH Terms: conditions — Melanoma; Neuroblastoma; Sarcoma; Osteosarcoma | interventions — lorukafusp alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DG2 positive relapsed or refractory solid tumors (Experimental): The initial hu14.18-IL2 fusion protein (FP) dose will be 2 mg/m2 given intravenously over 4 hours, daily for 3 days. Five separate dose levels are scheduled: 2 mg/m²/dose (IV over 4 hours) x 3 days, 4 mg/m²/dose (IV over 4 hours) x 3 days, 6 mg/m²/dose (IV over 4 hours) x 3 days, 8 mg/m²/dose (IV over 4 hours) x 3 days, 10 mg/m²/dose (IV over 4 hours) x 3 days.
  Interventions: Biological: hu14.18-IL2 fusion protein

INTERVENTIONS:
Biological: hu14.18-IL2 fusion protein

SUMMARY:
RATIONALE: Biological therapies such as hu14.18-interleukin-2 fusion protein use different ways to stimulate the immune system and stop cancer cells from growing.

PURPOSE: Phase I trial to study the effectiveness of hu14.18-interleukin-2 fusion protein in treating children who have refractory or recurrent neuroblastoma or other tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of hu14.18-interleukin-2 fusion protein in children with refractory or recurrent neuroblastoma or other GD2-positive tumors.
* Determine the toxicity and pharmacokinetics of the fusion protein in these patients.
* Determine the effect of the fusion protein on systemic immune modulation in these patients.
* Quantitate the antifusion protein antibodies in patients treated with fusion protein.
* Evaluate antitumor responses resulting from this fusion protein regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive hu14.18-interleukin-2 (hu14.18-IL2) fusion protein IV over 4 hours once daily on days 1-3. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of hu14.18-IL2 fusion protein until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 2 months for 1 year, every 6 months for 3 years, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 18-24 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed neuroblastoma or melanoma at original diagnosis

  * Refractory to chemotherapy or recurrence after prior multiagent chemotherapy
  * Measurable or evaluable (detectable by bone scan) metastatic disease OR
  * No evidence of disease if complete response to prior surgical resection, radiotherapy, and/or chemotherapy OR
* Histologically confirmed tumor expressing GD2 antigen at original diagnosis or relapse

  * Refractory to standard treatment
  * Measurable or evaluable disease by clinical assessments or laboratory markers OR
  * No evidence of disease after prior surgical resection of metastatic, recurrent disease
  * Histologically confirmed recurrent osteogenic sarcoma after prior chemotherapy allowed
  * Soft tissue sarcoma allowed
* No primary CNS tumors
* Prior CNS metastases allowed, provided:

  * Disease previously treated
  * Disease clinically stable for 4 weeks before study
  * At least 4 weeks since prior steroids for CNS metastases
* No clinically detectable pleural effusions or ascites

PATIENT CHARACTERISTICS:

Age:

* 21 and under

Performance status:

* Karnofsky 60-100% for children over age 10
* Lansky 60-100% for children age 10 and under

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count at least 75,000/mm^3 (transfusion allowed)
* Hemoglobin at least 9.0 g/dL (transfusion allowed)

Hepatic:

* Bilirubin less than 1.5 mg/dL
* ALT or AST no greater than 2.5 times normal
* Hepatitis B surface antigen negative

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance or radioisotope glomerular filtration rate at least 60 mL/min

Cardiovascular:

* Shortening fraction at least 27% by echocardiogram OR
* Ejection fraction more than 50% by MUGA scan
* No congestive heart failure
* No uncontrolled cardiac rhythm disturbance

Pulmonary:

* FEV_1 and FVC more than 60% of predicted OR
* No dyspnea at rest
* No exercise intolerance
* Oxygen saturation more than 94% by pulse oximetry on room air

Neurologic:

* No seizure disorders requiring antiseizure medications
* No significant neurologic deficit or grade 2 or greater objective peripheral neuropathy

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No significant concurrent illnesses unrelated to cancer or its treatment
* No significant psychiatric disabilities
* No uncontrolled active infections
* No uncontrolled active peptic ulcer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 week since prior growth factors
* At least 1 week since prior immunomodulatory therapy
* Prior monoclonal antibodies allowed if no detectable antibody to hu14.18
* Prior autologous bone marrow transplantation (BMT) or stem cell transplantation (SCT) allowed
* Prior autologous BMT or SCT with monoclonal antibody-purged specimens allowed
* No concurrent growth factors
* No concurrent interferon

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas, mitomycin, or melphalan)
* No concurrent palliative chemotherapy

Endocrine therapy:

* See Disease Characteristics
* At least 2 weeks since prior glucocorticoids, except for life-threatening symptoms
* No concurrent corticosteroids
* No concurrent glucocorticoids, except for life-threatening symptoms

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy
* No concurrent palliative radiotherapy

Surgery:

* See Disease Characteristics
* At least 2 weeks since prior major surgery (e.g., laparotomy or thoracotomy)
* No prior organ allografts
* No concurrent palliative surgery

Other:

* Recovered from prior therapy
* At least 1 week since prior tretinoin
* At least 3 weeks since prior immunosuppressive therapy
* No other concurrent immunosuppressive drugs

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2001-10; Primary Completion 2005-01 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Determine the MTD and pharmacokinetics of hu14.18-IL2 fusion protein
  Determine the MTD of hu14.18-IL2 fusion protein and determine the pharmacokinetics of the fusion protein when given as I.V. injections

SECONDARY OUTCOMES:
Assess immunological changes associated with fusion protein therapy

CONTACTS AND LOCATIONS:
Overall Officials: Paul M. Sondel, MD, PhD, Study Chair — University of Wisconsin, Madison
Locations (59):
- United States (54):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Shands Cancer Center at the University of Florida Health Science Center, Gainesville, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Scottish RiteCampus, Atlanta, Georgia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Kansas Cancer Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University Medical Center, St Louis, Missouri
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - University Hospital at State University of New York - Upstate Medical University, Syracuse, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Oklahoma University Medical Center at University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Texas Children's Cancer Center, Houston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (2):
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (3):
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec

REFERENCES:
- [Result] Osenga KL, Hank JA, Albertini MR, Gan J, Sternberg AG, Eickhoff J, Seeger RC, Matthay KK, Reynolds CP, Twist C, Krailo M, Adamson PC, Reisfeld RA, Gillies SD, Sondel PM; Children's Oncology Group. A phase I clinical trial of the hu14.18-IL2 (EMD 273063) as a treatment for children with refractory or recurrent neuroblastoma and melanoma: a study of the Children's Oncology Group. Clin Cancer Res. 2006 Mar 15;12(6):1750-9. doi: 10.1158/1078-0432.CCR-05-2000. PMID 16551859